CLINICAL TRIAL: NCT02899650
Title: Rates of Recovery From Strenuous Exercise in Physically Active Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a research project that was conducted by a visiting scholar and his time for departure came earlier than the study completion.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Hirofumi Tanaka, Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-04-0070
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Muscles
Keywords: Delayed Onset Muscle Soreness; Eccentric exercise; Masters athlete
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Young Fit (Experimental): Young (18-39 yrs) people who have endurance training habit
  Interventions: Other: exercise
- Young Unfit (Experimental): Young (18-39 yrs) people who have sedentary lifestyle.
  Interventions: Other: exercise
- Older Fit (Experimental): Older (50-80 yrs) people who have endurance training habit
  Interventions: Other: exercise
- Older Unfit (Experimental): Older (50-80 yrs) people who have sedentary lifestyle
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — acute downhill running

SUMMARY:
The purpose of this study to determine if older adults who are healthy and physically active (i.e., Masters athletes) demonstrate slower rates of recovery from unaccustomed strenuous exercise of downhill running than younger peers.

DETAILED DESCRIPTION:
There is a well-conceived notion that the recovery from strenuous exercise gets slower as individuals get older in age. Studies using animal models have demonstrated that stretching of electrically-activated skeletal muscle to mimic eccentric muscle contractions results in a greater decline and slower recovery in muscular force in old mice than in young mice. Similarly, in human studies using sedentary adults, age has been associated with a slower rate of recovery from a series of eccentric contractions. However, the process of aging is often confounded by coexisting diseases and gradual sedentary lifestyles that progress with advancing aging. Could older adults who are apparently healthy and habitually exercising demonstrate slower rates of recovery from strenuous exercise? In a small-scale study, recreationally-active middle-aged adults did not display a slower recovery from unaccustomed eccentric exercise than young adults. Masters athletes are an effective experimental model to address this question as extrinsic factors (e.g., deconditioning, chronic degenerative diseases) that often confound the intrinsic aging process can be minimized in this population. As no study has been conducted in Masters athletes, it is unknown if Masters athletes would experience slower rates of recovery similar to their sedentary peers.

With this information as background, the general aim of the proposed study is to determine if older adults who are healthy and physically active demonstrate slower rates of recovery from unaccustomed strenuous exercise of downhill running than younger peers. In an attempt to properly determine the influence of aging and regular physical activity, 4 groups of apparently healthy adults, including young sedentary, young trained, older sedentary, and older trained adults, will be studied.

A total of 60 apparently healthy men and women will serve as subjects. Half will be young [18-40-year-old (n=30)] and the other half older [50-80-year-old (n=30)]. After the screening and familiarization, investigators will ask participants to visit the laboratory four times (four consecutive days) to perform downhill running and to test physiological measurements (muscular strength, pain scale, range of motion, arterial stiffness and blood pressure and blood creatinine and myoglobin concentrations).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (exercise < 1 time/week) or well-trained individuals (exercise ≧ 2 times/week)
* Ages 18-39 and 50-80 years
* Individuals who can safely exercise

Exclusion Criteria:

* Individuals who reports "Symptoms or Signs Suggestive of Disease" on the Health Research Questionnaire (heart and respiratory problems, dizziness and ankle edema).
* Individuals who report substance abuse within the last 6 months (elicit drugs, alcohol)
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Lab at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavender AP, Nosaka K. Changes in markers of muscle damage of middle-aged and young men following eccentric exercise of the elbow flexors. J Sci Med Sport. 2008 Apr;11(2):124-31. doi: 10.1016/j.jsams.2006.11.004. Epub 2007 Mar 9. PMID 17350334
- [Background] Dedrick ME, Clarkson PM. The effects of eccentric exercise on motor performance in young and older women. Eur J Appl Physiol Occup Physiol. 1990;60(3):183-6. doi: 10.1007/BF00839156. PMID 2347319
- [Background] Brooks SV, Faulkner JA. Contraction-induced injury: recovery of skeletal muscles in young and old mice. Am J Physiol. 1990 Mar;258(3 Pt 1):C436-42. doi: 10.1152/ajpcell.1990.258.3.C436. PMID 2316632
- [Background] Brooks SV, Faulkner JA. The magnitude of the initial injury induced by stretches of maximally activated muscle fibres of mice and rats increases in old age. J Physiol. 1996 Dec 1;497 ( Pt 2)(Pt 2):573-80. doi: 10.1113/jphysiol.1996.sp021790. PMID 8961197
- See also: Pubmed — http://www.ncbi.nlm.nih.gov/pubmed

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We planned to recruit a total of 60 participants. However, we were not able to recruit older unfit adults so this group was dropped from the study. Additionally, this was a research project conducted by a visiting scholar and his departure approached quickly so the study was closed prematurely with smaller numbers in each group.
Period: Overall Study
Arm/Group | Young Fit | Young Unfit | Older Fit | Older Unfit
Started | 15 | 10 | 14 | 0 (We were not able to recruit older unfit adults so this group was dropped from the study.)
Completed | 15 | 10 | 14 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were not able to recruit older sedentary partcipants so this group was dropped from the data analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Fit | Young Unfit | Older Fit | Total
Number analyzed (Participants) | 15 | 10 | 14 | 39
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 27 (2) | 28 (2) | 58 (2) | 38 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 10 | 4 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 14 | 10 | 13 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Force Development
Description: Rate of force development are measured by determining peak torque achieved on an isometric leg extension machine.
Time Frame: After the downhill running protocol, various markers of muscle damage and muscular strength were obtained 24 hours post (the third visit), 48 hours post (the forth visit) and 72 hours post (the fifth visit).
Measure: Mean (Standard Error); unit: Nm
Arm/Group | Young Fit | Young Unfit | Older Fit
Number analyzed (Participants) | 15 | 10 | 14
Nm
  Baseline | 102 (3) | 108 (4) | 100 (2)
  24h post | 97 (3) | 106 (4) | 100 (3)
  48h post | 100 (2) | 106 (5) | 103 (3)
  72h post | 102 (2) | 105 (4) | 103 (2)

2. Secondary Outcome: Pain Scale
Description: Pain scale on quadriceps muscle was assessed using a validated visual pain scale. The scale was on a 10-point scale (0 being absence of soreness, 10 being worst imaginable soreness).
Time Frame: After the downhill running protocol, muscle damage pain scale was measured 24 hours post (the third visit), 48 hours post (the forth visit) and 72 hours post (the fifth visit).
Measure: Mean (Standard Error); unit: arbitrary scale unit from 0 to 10
Arm/Group | Young Fit | Young Unfit | Older Fit
Number analyzed (Participants) | 15 | 10 | 14
arbitrary scale unit from 0 to 10
  Baseline | 0.2 (0.1) | 0.1 (0.1) | 0.0 (0.0)
  24h post | 3.7 (0.5) | 4.7 (0.6) | 2.4 (0.6)
  48h post | 4.2 (0.6) | 4.9 (0.7) | 2.7 (0.6)
  72h post | 2.7 (0.5) | 3.2 (0.8) | 1.5 (0.4)

ADVERSE EVENTS:
Time Frame: Each participant was followed for a span of 4 days. After the downhill running protocol, various markers of muscle damage and muscular strength were obtained 24 hours post (the third visit), 48 hours post (the forth visit) and 72 hours post (the fifth visit).
Description: This is an acute exercise study. No adverse events were reported.
Arm/Group | Young Fit | Young Unfit | Older Fit | Older Unfit
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10 | 0/14 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/14 | 0/0
Other Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/14 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02899650/Prot_SAP_000.pdf